CLINICAL TRIAL: NCT01299636
Title: Phase I, Multicenter, Open-label, Dose-escalating, Clinical and Pharmacokinetic Study of PM060184 Administered Intravenously to Patients With Advanced Solid Tumors
Brief Title: Study of PM060184 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PM60184-A-002-10
Record Dates: First submitted 2011-02-09; First posted 2011-02-18 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Solid Tumors
Keywords: PM060184; Phase I; Pharma Mar
MeSH Terms: interventions — plocabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PM060184 (Experimental)
  Interventions: Drug: PM060184

INTERVENTIONS:
Drug: PM060184 — PM060184 administered intravenously (i.v.) over 10 minutes at a starting dose of 4 mg/m2/day on three consecutive days q2w (on Days 1-3 and 15-17) every 28 days.

SUMMARY:
The purpose of the study is to determine the maximum tolerated dose and the recommended dose and to evaluate the safety and tolerability of PM060184.

DETAILED DESCRIPTION:
This trial intends to determine the maximum tolerated dose and the recommended dose, to evaluate the safety and tolerability, to determine the pharmacokinetics and to evaluate the antitumor activity of PM060184 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion criteria

1. Voluntary signed and dated written informed consent.
2. Patients with advanced solid tumors refractory to Standard therapy.
3. Age >/= 18 years.
4. Recovery from drug-related adverse events (AEs) of previous treatments, excluding alopecia.
5. Normal laboratory values within seven days prior to treatment administration.
6. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both men and women must agree to use a medically acceptable method of contraception throughout the treatment period and for three months after discontinuation of treatment.

Exclusion criteria

1. Pregnant or lactating women.
2. Less than three weeks from radiation therapy or last dose of hormonal therapy, biological therapy or chemotherapy
3. Prior treatment with any investigational product less than 30 days prior to the first.
4. Central Nervous System metastases
5. Other relevant diseases or adverse clinical conditions:

   * Increased cardiac risk:
   * Presence of significant neurological or psychiatric disorders
   * Neuropathy
   * Active infection requiring treatment.
   * Liver disease (e.g., cirrhosis, hepatitis).
   * Immunocompromised patients.
   * Any other major illness.
6. Limitation of the patient's ability to comply with the treatment.
7. Known hypersensitivity to any of the components of the drug product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
MTD (maximum tolerated dose) and RD (recommended dose) of PM060184. | From treatment onset to end of treatment
  To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM060184 administered on Days 1 and 8 of a 21-day cycle intravenously (i.v.) over 10 minutes to patients with advanced solid tumors.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of this drug in patients who have advanced solid tumors. | Blood samples will be collected up to 48 hours after the first infusion. At the RD, 24-h urine collection samples and 15 additional blood samples up to 48 hours after the second infusion of the first cycle.
  The complete plasma concentration-time profiles of PM06184 will be analyzed by standard non-compartmental methods.The percent of PM060184 total dose excreted unchanged into the urine over the collection interval will be calculated from the urine samples.
Antitumor activity | Every six weeks while on treatment. Patients who discontinued treatment without disease progression will be followed every three months until disease progression, other antitumor therapy, death or until the end-of-study date, whichever occurs first.
  Antitumor activity will be measured according to the RECIST (Response Evaluation Criteria In Solid Tumors) version 1.1 or by evaluation of tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Papadopoulos, MD, Principal Investigator — START- South Texas Accelerated Research Therapeutics, LLC
Locations (1):
- START- South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas, United States